CLINICAL TRIAL: NCT05878236
Title: iMmune SignAtures and Clinical outComes in Acute Pancreatitis: the MoSAIC Study
Brief Title: iMmune SignAtures and Clinical outComes in AP
Acronym: MoSAIC
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: University of Pittsburgh (Other); University of Illinois at Chicago (Other); University of Southern California (Other); Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, George Papachristou, Professor of Internal Medicine, Director of Gastroenterology, Ohio State University
Other Study IDs: 2022H0394
Record Dates: First submitted 2023-03-20; First posted 2023-05-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Pancreatitis
Keywords: Acute Pancreatitis; Immunology; MoSAIC
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy Coat from Plasma samples will be collected and stored for genetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute Pancreatitis: Patients meeting Revised Atlanta Criteria for diagnosis of acute pancreatitis
  Interventions: Diagnostic Test: CyTOF Analysis

INTERVENTIONS:
Diagnostic Test: CyTOF Analysis — CyTOF laboratory testing for cytokine levels to correlate with severity of acute pancreatitis

SUMMARY:
The MoSAIC study is a prospective, observational study designed to develop an early prediction tool for severe acute pancreatitis (SAP) and define a distinct immunologic profile compared to moderate acute pancreatitis (MAP). The aims are to validate a new multi-cytokine panel for early prediction of SAP and to identify the specific immune cells that correspond with cytokine signatures in early acute pancreatitis to characterize the immune pathways driving the development of SAP. Participants will provide blood samples and complete patient surveys and interviews within 36 hours of hospital presentation, at 48 hours, and hospital day 7 (if admitted). Data on hospital stay, medical history, clinical course, and severity of disease will be collected.

DETAILED DESCRIPTION:
All participants will sign an informed consent before participating in the study. Adult subjects of both sexes and belonging to all ethnicities will be enrolled. Participants will consent for access to their electronic health records, complete study questionnaires, undergo serial clinical laboratory testing and provide biospecimens during their acute pancreatitis (AP) hospitalization. The research team will access the electronic health records for 5 years from the time of enrollment in the study.

The study network is comprised of five academic sites. Four sites will enroll AP patients [OSU, University of Illinois in Chicago Hospital (UIC), University of Pittsburgh Medical Center (UPMC), and the Keck Hospital of the University of Southern California (USC)]. The fifth site, the Benaroya Research Institute (BRI) will coordinate biospecimen handling for analyses, perform bioinformatics and serve as the biospecimen coordinating center (BCC). Each enrolling site will collect and ship biosamples to BRI. The blood samples collected in this study will be deposited into the Benaroya Research Institute (BRI) Immune-Mediated Diseases Registry and Repository (IMDRR). Participation in the repository is a requirement for inclusion in the study. Specimens collected in this study will be used for immune assays. Samples will also be coded and stored for up to 15 years in the IMDRR. Samples may be used to evaluate additional responses as new research tools become available or exploratory hypotheses are generated. OSU will serve as the data coordinating center (DCC). Coordinators at enrolling sites will enter study data into a secure cloud-based electronic database, and the DCC will be in charge of monitoring the quality and completeness of the electronic data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years at the time of enrollment
2. Diagnosis of acute pancreatitis (AP) according to the revised Atlanta criteria (see definition below)
3. Participant is approached by the research team within 36 hours of presentation to the hospital
4. Participant fully understands and agrees to participate in all aspects of the study, including providing informed consent, completion of interviews and data forms, and collection of biospecimens

Acute pancreatitis is defined/diagnosed using the revised Atlanta criteria, which requires the presence of at least two of the following criteria:

i. Upper abdominal pain ii. Elevation of serum amylase or lipase level to >/=3 times the upper limit of normal iii. Features of AP on cross-sectional imaging.

Exclusion Criteria:

1. Diagnosis of definite chronic pancreatitis (CP) at enrollment (see also study definitions) based on either of the following criteria met by computed tomography (CT) scan (including non-contrast enhanced) or Magnetic resonance Imaging (MRI) or Magnetic Resonance Cholangiopancreatography (MRCP):

   i. Parenchymal or ductal calcifications on CT scan (after excluding the possibility that calcifications are vascular) ii. Intraductal filling defects suggestive of calcifications on MRI and/or MRCP iii. Non-contrast imaging is acceptable for the assessment of definite CP, but calcifications noted by endoscopic ultrasound only (and not correlated with CT) are not considered definite CP. Patients with autoimmune pancreatitis, but no evidence of calcifications, may still be enrolled, assuming they satisfy inclusion criteria for 'diagnosis of AP'
2. Potential participants with post-ERCP AP who are expected to be hospitalized for less than 48 hours.
3. Pancreatic tumors, including ductal adenocarcinoma, neuroendocrine tumors, and metastasis.
4. Confirmed or suspected cystic tumor associated with main pancreatic duct dilation or believed to be the cause of AP (in the site-PI's judgment).
5. Prior pancreatic surgery, including, but not limited to distal pancreatectomy, pancreaticoduodenectomy, pancreatic necrosectomy, and Frey procedure.
6. Severe systemic illness that in the judgment of the investigative team will confound outcome assessments and immunological outcomes or pose additional risk for harm, including the history of solid organ transplant, acquired immunodeficiency syndrome (AIDS), active treatment for cancer (except non-melanoma skin cancer) within 12 months prior to enrollment, chronic kidney disease with eGFR <30 or on dialysis prior to AP, and cirrhosis (based on imaging or biopsy), or any other medical condition that in the opinion of the site-PI carries a life expectancy of <12 months.
7. Known pregnancy at the time of enrollment.
8. Incarceration.
9. Any other condition or factor that would compromise the participant's safety or the scientific integrity of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who meet all inclusion and no exclusion criteria will be considered for enrollment. Patients presenting to the hospital or emergency room with acute pancreatitis (AP) will be screened and enrolled within 36 hours of presentation to capture relevant biomarker information as early in their episode of AP as possible. Patients with chronic calcific pancreatitis, severe systemic illness confounding severity assessments or immunological outcomes, or anyone with an altered or compromised immune system will be excluded from enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Multi-Cytokine Panel Validation | 4 years
  Validate a novel multi-cytokine panel for early prediction of severe acute pancreatitis. The panel includes IL-8, TNFa R1, HGF, Resistin and Angiopoietin-2.
Cytokine Signature Correlation | 4 years
  Correlate temporal cytokine signatures with disease severity. We will be correlating the above cytokines as well Il-6 and MCP-1.

SECONDARY OUTCOMES:
Circulating Immune Cells | 4 years
  Identify circulating immune cells that correspond with cytokine signatures in early acute pancreatitis
Immune Pathways | 4 years
  Characterize the immune pathways driving the development of severe acute pancreatitis

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - University of Illinois Chicago, Chicago, Illinois
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided